CLINICAL TRIAL: NCT05355506
Title: National Taipei University of Nursing and Science
Brief Title: The Development and Effectiveness of Heart Failure Self-Health Management Application
Acronym: APP
Status: Suspended | Type: Observational
Why Stopped: covid-19
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Assistant Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: 19MMHIS04Oe
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Development and Effectiveness of Heart Failure Self-Health Management Application: Heart Failure can cause physical disability and death. According to the Ministry of Health and Welfare, there were 20,644 deaths from heart disease, ranking second among the top 10 causes of death [1]. The World Health Organization (WHO) has advocated nursing guidance with the concept of "empowerment", where patients can play an active and aggressive role in managing their health [2]. This paperless nursing health education guidance information can be designed through the application, which features non-professional expressions and visualization methods. The users can participate in feedback-based interactions and complete the questionnaires after receiving nursing guidance. This study used the Technology Acceptance Model (TAM) to evaluate patients' acceptance of the nursing guidance application and the effectiveness of such nursing guidance.
  Interventions: Device: Application

INTERVENTIONS:
Device: Application — Knowledge & record

SUMMARY:
Aims: To develop a smartphone application and investigate its effectiveness on patients with heart failure after using the "heart failure self-health management application.".

DETAILED DESCRIPTION:
Abstract Aims: To develop a smartphone application and investigate its effectiveness on patients with heart failure after using the "heart failure self-health management application.".

Design: The single-group pre- and post-test experimental design was adopted. Methods: This study used convenience sampling and the one-group pretest and posttest design as the research methods and developed the "heart failure self-health management application" using the Google cloud database and Web App. The research period was from July 1 to December 31, 2019, a total of 36 patients diagnosed with heart failure during hospitalization completed the pretest and posttest. This App (1) provides text and video heart failure self-care knowledge content; (2) enables users to record and browse blood pressure, heart rate, and weight; and (3) provides the data from the Dutch Heart Failure Knowledge Scale and Technology Acceptance Model.

Keywords: heart failure; self-health management; application

ELIGIBILITY:
Inclusion Criteria:

* Heart failure

Exclusion Criteria:

* Health

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Heart failure
  Exclusion Criteria:
  * Health
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-03 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
participant's knowledge about heart failure significantly increased after the intervention | 6 months
  Provides the data from the Dutch Heart Failure Knowledge Scale and Technology Acceptance Model. Analysis on participant's knowledge about heart failure and Technology Acceptance Model Scale after the Intervention. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Pei-Hung Liao, Taipei County, Taiwan